CLINICAL TRIAL: NCT04575948
Title: Antibacterial, Antiplaque and Anticariogenic Effect of Moringa Oleifera Mouthwash Compared to Chlorhexidine Mouthwash: A Randomized Clinical Trial
Brief Title: Anticariogenic Effect of Moringa Oleifera Mouthwash Compared to Chlorhexidine Mouthwash
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Misr International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PER8273010
Record Dates: First submitted 2020-09-23; First posted 2020-10-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-03

CONDITIONS: Plaque, Dental; Antimicrobial; Mouthwash; Cytotoxicity
Keywords: Moringa Oleifera; antibacterial activity; mouthwash; chlorhexidine; antiplaque; herbal; translational research
MeSH Terms: conditions — Dental Plaque | interventions — flocculant protein MO 2.1, Moringa oleifera; hexitol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Masking of all caregivers, examiners (I) and (II), as well as patients are planned. No one other than HSE at the NRC will know which mouthwash is in each bottle. HSE will not be involved in patient recruitment, follow-up or assessment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moringa Oleifera mouth wash (Experimental): According to part I of the study, we will select the most effective (Non-toxic, anti-bacterial effect) Moringa extract to prepare the mouth wash.
  Interventions: Drug: Moringa Oleifera
- Base formula of mouth wash (Placebo Comparator): Base formula of mouthwash
  Interventions: Drug: Base formula
- Chlorhexidine (Active Comparator): Commercial 0.12% chlorhexidine digluconate mouthwash
  Interventions: Drug: Chlorhexidine mouthwash

INTERVENTIONS:
Drug: Moringa Oleifera — Non toxic Moringa extract with antibacterial and antiplaque effect will be used
  Arms: Moringa Oleifera mouth wash
Drug: Chlorhexidine mouthwash — Commercial 0.12% chlorhexidine digluconate mouthwash twice daily (each morning and before bedtime during the 21-day study period) after intake of food. The patient will be asked to use 15 ml of mouthwash swish it for 60 sec. then expectorate.
  Other Names: Hexitol
  Arms: Chlorhexidine
Drug: Base formula — Base formula is a negative control
  Arms: Base formula of mouth wash

SUMMARY:
Moringa oleifera (MO) is an extraordinary nutritious vegetable tree with high medicinal value for its antibacterial properties. Formulation of various natural dental remedies from this plant and their testing for their effectiveness might yield promising antibacterial, antiplaque and anticariogenic agents with minimal side effects.

Aim of the study:

Part I: The aim of this in-vitro part of the study is to formulate a nontoxic mouthwash from MO leaves extract, having antimicrobial activity, to be used in part II of the study. Furthermore, stability and efficacy of the developed mouth wash will be evaluated.

Part II: The aim of this randomized controlled trial is to evaluate the antibacterial, antiplaque and anticariogenic effect of MO mouthwash compared to chlorhexidine mouthwash.

DETAILED DESCRIPTION:
Statement of the problem: Oral diseases remain a major health problem all over the world. Periodontal diseases and dental caries are the most common non-communicable oral diseases in mankind and the leading cause of tooth loss. Both diseases can lead to nutritional compromise and negative impact on self-esteem and quality of life. As the International situation is now changing towards the use of non- toxic and environmentally friendly products, development of modern drugs from traditional medicinal plants should be emphasized for the control of various human diseases. Moringa oleifera (MO) is an extraordinary nutritious vegetable tree with high medicinal value for its antibacterial properties. Formulation of various natural dental remedies from this plant and their testing for their effectiveness might yield promising antibacterial, antiplaque and anticariogenic agents with minimal side effects.

Aim of the study:

Part I: The aim of this in-vitro part of the study is to formulate a nontoxic mouthwash from MO leaves extract, having antimicrobial activity, to be used in part II of the study. Furthermore, stability and efficacy of the developed mouth wash will be evaluated.

Part II: The aim of this randomized controlled trial is to evaluate the antibacterial, antiplaque and anticariogenic effect of MO mouthwash compared to chlorhexidine mouthwash.

Materials and Methods:

Part I: In this part of the study; MO leaves will be extracted using different solvents. The active constituents in the form of total phenolic content (TPC) and total flavonoid content (TFC) of the developed extract will be assayed. All the prepared extracts will be evaluated for their antibacterial activity against S. mutans and P. gingivalis. The MO extract(s), which have the highest antibacterial activity will be tested for the cytotoxicity effect on gingival fibroblast cells using cell culture facilities and MTT [3-(4, 5-dimethylthiazol-2-yl)-2, 5-diphenyl tetrazolium bromide] assay. The MO mouth wash will be prepared after determination of the minimum inhibitory concentration (MIC) for the extract with the highest antibacterial activity and non-cytotoxic effect. Eventually stability and efficacy of the developed mouth wash will be tested under different storage conditions.

Part II: A triple-blind, parallel arm, randomized controlled clinical trial involving 90 patients with biofilm-induced gingivitis (plaque-induced gingivitis) and moderate-high caries risk will be carried out. Patients will be divided equally into three groups and will receive either the base formula mouthwash (BF; negative control), MO incorporated into the base formula mouthwash or commercial 0.12% Chlorhexidine HCL mouthwash (Hexitol®, H; positive control). After professional oral prophylaxis (scaling and polishing), clinical parameters measurement (gingival index, plaque index, modified sulcular bleeding index, stain index) will be determined for the project. Unstimulated saliva and plaque samples for Streptococcus mutans colony forming units (CFU) will be collected at baseline, 7th, 14th and 21st days. Salivary flow, salivary pH and International Caries Detection and Assessment System II (ICDAS II), will be recorded at baseline, 21st day, 3 months and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Systemically free as reported by the patients
* Minimum of 20 teeth present in the dentition (excluding wisdom teeth);
* Clinically healthy gingiva (on intact periodontium)
* Dental biofilm-induced gingivitis (plaque induced gingivitis) according to the criteria set by the American Academy of Periodontology for classification of periodontal diseases and conditions in 2017
* Moderate to high caries risk patients

Exclusion Criteria:

* Patients with periodontitis or requiring other immediate dental treatments (within the current 6 months)
* Subjects on antibiotics within last 6 months
* Periodontal therapy for the past 6 months
* Pregnant women and lactating mothers
* Medically compromised patients
* Subjects with tobacco consumption in any form
* Subjects wearing partial dentures or having clinically unacceptable restorations or bridges
* Subjects wearing orthodontic appliances
* History of allergy to chemical or any herbal products

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2027-12 (Estimated); Primary Completion 2028-11 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Gingival index (GI) | 21 days
  as assessed by Lӧe and Silness: Score from 0 to 3, Zero is normal subject
White Spot Lesions | 21 days
  Assessed by ICDAS II: Scores from 0 to 9: Zero is unrestored or unsealed tooth surface

CONTACTS AND LOCATIONS:
Overall Officials: Mahassen M Farghaly, Professor, Study Chair — Vice president of community services and environmental awareness

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsh PD. Dental plaque as a microbial biofilm. Caries Res. 2004 May-Jun;38(3):204-11. doi: 10.1159/000077756. PMID 15153690
- [Background] Marsh PD, Martin MV. Oral microbiology. 5th edition. Edinburgh (UK): Churchil Livingstone; 2009. P 92-110
- [Background] Tanzer JM, Livingston J, Thompson AM. The microbiology of primary dental caries in humans. J Dent Educ. 2001 Oct;65(10):1028-37. PMID 11699974
- [Background] Loesche WJ. Role of Streptococcus mutans in human dental decay. Microbiol Rev. 1986 Dec;50(4):353-80. doi: 10.1128/mr.50.4.353-380.1986. No abstract available. PMID 3540569
- [Background] Marsh PD, Nyvad B. The oral microflora and biofilms on teeth. In: Fejerskov O, Kidd E, editors. Dental caries. The disease and its clinical management. 2nd edition. Oxford: Blackwell; 2008. p. 163-87.
- [Background] Marsh PD. Microbiology of dental plaque biofilms and their role in oral health and caries. Dent Clin North Am. 2010 Jul;54(3):441-54. doi: 10.1016/j.cden.2010.03.002. PMID 20630188
- [Background] Silverstone LM, Hicks MJ, Featherstone MJ. Dynamic factors affecting lesion initiation and progression in human dental enamel. Part I. The dynamic nature of enamel caries. Quintessence Int. 1988 Oct;19(10):683-711. No abstract available. PMID 3269557
- [Background] Al-Obaidi R, Salehi H, Desoutter A, Bonnet L, Etienne P, Terrer E, Jacquot B, Levallois B, Tassery H, Cuisinier FJG. Chemical & Nano-mechanical Study of Artificial Human Enamel Subsurface Lesions. Sci Rep. 2018 Mar 6;8(1):4047. doi: 10.1038/s41598-018-22459-7. PMID 29511281
- [Background] Mini KJ, Anulekh B, Anupama G. Incipient caries: an early intervention approach. Int J Community Med Public Health 2015; 2(1):10-14
- [Background] Wennerholm K, Lindquist B, Emilson CG. The toothpick method in relation to other plaque sampling techniques for evaluating mutans streptococci. Eur J Oral Sci. 1995 Feb;103(1):36-41. doi: 10.1111/j.1600-0722.1995.tb00008.x. PMID 7600248
- [Background] Dasanayake AP, Caufield PW, Cutter GR, Roseman JM, Kohler B. Differences in the detection and enumeration of mutans streptococci due to differences in methods. Arch Oral Biol. 1995 Apr;40(4):345-51. doi: 10.1016/0003-9969(94)00164-7. PMID 7605262
- [Background] Pitts N. "ICDAS"--an international system for caries detection and assessment being developed to facilitate caries epidemiology, research and appropriate clinical management. Community Dent Health. 2004 Sep;21(3):193-8. No abstract available. PMID 15470828
- [Background] Ismail AI, Sohn W, Tellez M, Amaya A, Sen A, Hasson H, Pitts NB. The International Caries Detection and Assessment System (ICDAS): an integrated system for measuring dental caries. Community Dent Oral Epidemiol. 2007 Jun;35(3):170-8. doi: 10.1111/j.1600-0528.2007.00347.x. PMID 17518963
- [Background] Braga MM, Oliveira LB, Bonini GA, Bonecker M, Mendes FM. Feasibility of the International Caries Detection and Assessment System (ICDAS-II) in epidemiological surveys and comparability with standard World Health Organization criteria. Caries Res. 2009;43(4):245-9. doi: 10.1159/000217855. Epub 2009 May 8. PMID 19439944
- [Background] Almosa NA, Lundgren T, Bresin A, Birkhed D, Kjellberg H. Diagnosing the severity of buccal caries lesions in orthodontic patients at de-bonding using digital photographs. Acta Odontol Scand. 2014 Aug;72(6):474-80. doi: 10.3109/00016357.2013.865788. Epub 2013 Dec 9. PMID 24320004
- [Background] Preus HR, Aass AM, Hansen BF, Moe B, Gjermo P. A randomized, single-blind, parallel-group clinical study to evaluate the effect of soluble beta-1,3/1,6-glucan on experimental gingivitis in man. J Clin Periodontol. 2008 Mar;35(3):236-41. doi: 10.1111/j.1600-051X.2007.01183.x. PMID 18269662
- [Background] LOE H, THEILADE E, JENSEN SB. EXPERIMENTAL GINGIVITIS IN MAN. J Periodontol (1930). 1965 May-Jun;36:177-87. doi: 10.1902/jop.1965.36.3.177. No abstract available. PMID 14296927
- [Background] Theilade E, Wright WH, Jensen SB, Loe H. Experimental gingivitis in man. II. A longitudinal clinical and bacteriological investigation. J Periodontal Res. 1966;1:1-13. doi: 10.1111/j.1600-0765.1966.tb01842.x. No abstract available. PMID 4224181
- [Background] Cobb CM. Non-surgical pocket therapy: mechanical. Ann Periodontol. 1996 Nov;1(1):443-90. doi: 10.1902/annals.1996.1.1.443. No abstract available. PMID 9118268
- [Background] Pradeep AR, Suke DK, Martande SS, Singh SP, Nagpal K, Naik SB. Triphala, a New Herbal Mouthwash for the Treatment of Gingivitis: A Randomized Controlled Clinical Trial. J Periodontol. 2016 Nov;87(11):1352-1359. doi: 10.1902/jop.2016.130406. Epub 2016 Jul 21. PMID 27442086
- [Background] Budtz-Jorgensen E, Loe H. Chlorhexidine as a denture disinfectant in the treatment of denture stomatitis. Scand J Dent Res. 1972;80(6):457-64. doi: 10.1111/j.1600-0722.1972.tb00314.x. No abstract available. PMID 4575037
- [Background] Manipal S, Hussain S, Wadgave U, Duraiswamy P, Ravi K. The Mouthwash War - Chlorhexidine vs. Herbal Mouth Rinses: A Meta-Analysis. J Clin Diagn Res. 2016 May;10(5):ZC81-3. doi: 10.7860/JCDR/2016/16578.7815. Epub 2016 May 1. PMID 27437366
- [Background] Charles CH, Mostler KM, Bartels LL, Mankodi SM. Comparative antiplaque and antigingivitis effectiveness of a chlorhexidine and an essential oil mouthrinse: 6-month clinical trial. J Clin Periodontol. 2004 Oct;31(10):878-84. doi: 10.1111/j.1600-051X.2004.00578.x. PMID 15367192
- [Background] Rath SK, Singh M. Comparative clinical and microbiological efficacy of mouthwashes containing 0.2% and 0.12% chlorhexidine. Dent Res J (Isfahan). 2013 May;10(3):364-9. PMID 24019806
- [Background] Ruiz-Linares M, Ferrer-Luque CM, Arias-Moliz T, de Castro P, Aguado B, Baca P. Antimicrobial activity of alexidine, chlorhexidine and cetrimide against Streptococcus mutans biofilm. Ann Clin Microbiol Antimicrob. 2014 Aug 20;13:41. doi: 10.1186/s12941-014-0041-5. PMID 25139679
- [Background] Fischman SL. The history of oral hygiene products: how far have we come in 6000 years? Periodontol 2000. 1997 Oct;15:7-14. doi: 10.1111/j.1600-0757.1997.tb00099.x. PMID 9643227
- [Background] Abd Rani NZ, Husain K, Kumolosasi E. Moringa Genus: A Review of Phytochemistry and Pharmacology. Front Pharmacol. 2018 Feb 16;9:108. doi: 10.3389/fphar.2018.00108. eCollection 2018. PMID 29503616
- [Background] Khawaja TM, Tahira M, Ikram UK. Moringa oleifera: a natural gift - A review. J Pharm Sci Res. 2010; 2:775-81
- [Background] Mehta K, Balaraman R, Amin AH, Bafna PA, Gulati OD. Effect of fruits of Moringa oleifera on the lipid profile of normal and hypercholesterolaemic rabbits. J Ethnopharmacol. 2003 Jun;86(2-3):191-5. doi: 10.1016/s0378-8741(03)00075-8. PMID 12738086
- [Background] Fahey W. J. (2005). Moringa oleifera: a review of the medical evidence for its nutritional, therapeutic, and prophylactic properties. Part 1. Trees Life J. 1, 1-24
- [Background] Farooq, F., M. Rai, A. Tiwari, A. Khan, S. Farooq. Medicinal properties of Moringa oleifera: An overview of promising healer. J. of Medicinal Plants Research, 2012; 6(27): 4368-4374
- [Background] Mahdi, HarithJameel & Yousif, EmadMuthana & Khan, NurzalinaAbdulKarim & Mahmud, Roziahanim & Murugaiyah, Vikneswaran & Asmawi, Mohd. (2016). OPTIMIZING EXTRACTION CONDITIONS OF MORINGA OLEIFERA LAM LEAF FOR PERCENT YIELD, TOTAL PHENOLICS CONTENT, TOTAL FLAVONOIDS CONTENT AND TOTAL RADICAL SCAVENGING ACTIVITY.. International Journal of Advanced Research. 4. 682-695. 10.21474/IJAR01/2133.
- [Background] Caceres A, Cabrera O, Morales O, Mollinedo P, Mendia P. Pharmacological properties of Moringa oleifera. 1: Preliminary screening for antimicrobial activity. J Ethnopharmacol. 1991 Jul;33(3):213-6. doi: 10.1016/0378-8741(91)90078-r. PMID 1921416
- [Background] Abdull Razis AF, Ibrahim MD, Kntayya SB. Health benefits of Moringa oleifera. Asian Pac J Cancer Prev. 2014;15(20):8571-6. doi: 10.7314/apjcp.2014.15.20.8571. PMID 25374169
- [Background] Elgamily H, Moussa A, Elboraey A, El-Sayed H, Al-Moghazy M, Abdalla A. Microbiological Assessment of Moringa Oleifera Extracts and Its Incorporation in Novel Dental Remedies against Some Oral Pathogens. Open Access Maced J Med Sci. 2016 Dec 15;4(4):585-590. doi: 10.3889/oamjms.2016.132. Epub 2016 Nov 28. PMID 28028395
- [Background] Fajriani MS, Intania N. Effectiveness of Gargle with extract of leaf moringa (Moringa Oleifera)to plaque formation for ECC (Early Childhood Caries). Journal of Baghdad college of dentistry 2018; 23(2): 110-113
- [Background] Hartoyo M, Purnomo SE , Budiyati , Lestari KP, Sawab. The Effect of Mouth washing with Moringa Olivera to acidity saliva level of Diabetes Mellitus Patients. JMSCR 2017 ; 5(12): 32092-32096
- [Background] Pithon MM, Sant'Anna LI, Baiao FC, dos Santos RL, Coqueiro Rda S, Maia LC. Assessment of the effectiveness of mouthwashes in reducing cariogenic biofilm in orthodontic patients: a systematic review. J Dent. 2015 Mar;43(3):297-308. doi: 10.1016/j.jdent.2014.12.010. Epub 2015 Jan 6. PMID 25572792
- [Background] LOE H, SILNESS J. PERIODONTAL DISEASE IN PREGNANCY. I. PREVALENCE AND SEVERITY. Acta Odontol Scand. 1963 Dec;21:533-51. doi: 10.3109/00016356309011240. No abstract available. PMID 14121956
- [Background] Marsh PD, Nyvad B. The oral microflora and biofilms on teeth. In: Fejerskov O, Kidd E, editors. Dental caries. The disease and its clinical management. 2nd edition. Oxford: Blackwell; 2008. p. 163-87
- [Background] Zhao B. , Deng J, Li H, Yaqiang He, Tao Lan, Di Wu, Haodi Gong, Yan Zhang, and Zhicheng Chen , Optimization of Phenolic Compound Extraction from Chinese Moringa oleifera Leaves and Antioxidant Activities Beibei , Journal of Food Quality. 2019; 2019:1-14
- [Background] Seleshe S, Kang SN. In Vitro Antimicrobial Activity of Different Solvent Extracts from Moringa stenopetala Leaves. Prev Nutr Food Sci. 2019 Mar;24(1):70-74. doi: 10.3746/pnf.2019.24.1.70. Epub 2019 Mar 31. PMID 31008099
- [Background] Vermerie N, Malbrunot C, Azar M, Arnaud P. Stability of nystatin in mouthrinses; effect of pH temperature, concentration and colloidal silver addition, studied using an in vitro antifungal activity. Pharm World Sci. 1997 Aug;19(4):197-201. doi: 10.1023/a:1008664917377. PMID 9297733
- [Background] Murakami S, Mealey BL, Mariotti A, Chapple ILC. Dental plaque-induced gingival conditions. J Periodontol. 2018 Jun;89 Suppl 1:S17-S27. doi: 10.1002/JPER.17-0095. PMID 29926958
- [Background] Sanchez-Perez L, Acosta-Gio AE, Mendez-Ramirez I. A cluster analysis model for caries risk assessment. Arch Oral Biol. 2004 Sep;49(9):719-25. doi: 10.1016/j.archoralbio.2004.02.012. PMID 15275859
- [Background] Hefti AF, Preshaw PM. Examiner alignment and assessment in clinical periodontal research. Periodontol 2000. 2012 Jun;59(1):41-60. doi: 10.1111/j.1600-0757.2011.00436.x. PMID 22507059
- [Background] Chitharanjan S, Mithra N, Darshana D. Correlation between dental caries with salivary flow, pH, and buffering capacity in adult South Indian population: an in vivo study. Int. J. Res. Ayurveda Pharm 2013; 4(2): 219-223
- [Background] Sakeenabi B, Hiremath SS. Dental caries experience and salivary Streptococcus mutans, lactobacilli scores, salivary flow rate, and salivary buffering capacity among 6-year-old Indian school children. J Int Soc Prev Community Dent. 2011 Jul;1(2):45-51. doi: 10.4103/2231-0762.97697. PMID 24478953
- [Background] Lindquist B, Emilson CG. Dental location of Streptococcus mutans and Streptococcus sobrinus in humans harboring both species. Caries Res. 1991;25(2):146-52. doi: 10.1159/000261358. PMID 2059977
- [Background] SILNESS J, LOE H. PERIODONTAL DISEASE IN PREGNANCY. II. CORRELATION BETWEEN ORAL HYGIENE AND PERIODONTAL CONDTION. Acta Odontol Scand. 1964 Feb;22:121-35. doi: 10.3109/00016356408993968. No abstract available. PMID 14158464
- [Background] Lobene RR. Effect of dentifrices on tooth stains with controlled brushing. J Am Dent Assoc. 1968 Oct;77(4):849-55. doi: 10.14219/jada.archive.1968.0298. No abstract available. PMID 5244497
- [Background] Ainamo J, Bay I. Problems and proposals for recording gingivitis and plaque. Int Dent J. 1975 Dec;25(4):229-35. PMID 1058834